CLINICAL TRIAL: NCT00482404
Title: Study of the Effects of Romantic Affection on Blood Lipids, Blood Glucose, C-Reactive Protein, and Antibodies to Latent Epstein-Barr Virus
Brief Title: Effects of Romantic Affection on Blood Chemistry and Immune Parameters
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Arizona State University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1001 R03 MH075757-01A1
Record Dates: First submitted 2007-06-04; First posted 2007-06-05 (Estimated); Last update posted 2007-06-05 (Estimated); Status verified 2007-06

CONDITIONS: Stress; Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Romantic kissing

SUMMARY:
This trial tests the hypothesis that increasing nonverbal affection in romantic relationships will improve blood lipid parameters (total cholesterol, high and low density lipoproteins, triglycerides), blood glucose, and immune parameters (C-reactive protein and antibodies to latent Epstein-Barr virus). 52 healthy cohabiting romantic couples took part. In half of the couples, one partner increased the frequency of romantic kissing with the other partner during the six-week trial. The other couples received no such instruction. Blood tests performed before and after the trial were used to assess the health outcomes.

ELIGIBILITY:
Inclusion Criteria:

* 18+ years of age;
* English-speaking;
* Current co-habitation with romantic partner

Exclusion Criteria:

* History of hypercholesterolemia;
* Current pregnancy;
* Current use of blood-thinning agents;
* Greater than moderate anxiety about giving capillary blood;
* Weight of less than 110 pounds

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Dates: Start 2007-02; Study Completion 2007-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kory Floyd, PhD, Principal Investigator — Arizona State University